CLINICAL TRIAL: NCT02030054
Title: Pharmacodynamic Comparison of Rosuvastatin Versus Atorvastatin on Platelet Reactivity in Patients With Coronary Artery Disease on Dual Antiplatelet Therapy With New P2Y12 Inhibitors
Brief Title: Pharmacodynamic Comparison of Rosuvastatin Versus Atorvastatin on Platelet Reactivity in Patients With Coronary Artery Disease on Dual Antiplatelet Therapy With New P2Y12 Inhibitors (Trial gRANADa)
Acronym: gRANADa
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Polacco Marina, MD, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060114
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- atorvastatin (Active Comparator): Patients were randomly assigned to atorvastatin (40 mg day) or rosuvastatin (20 mg day) for 30 days. After 1-week wash-out period to avoid any carryover effect, cross-over was performed, and patients were switched to the other drug which was continued for 30 days.
  Interventions: Drug: Atorvastatin; Drug: Rosuvastatin
- rosuvastatin (Active Comparator): Patients were randomly assigned to atorvastatin (40 mg day) or rosuvastatin(20 mg day) for 30 days. After 1-week wash-out period to avoid any carryover effect, cross-over was performed, and patients were switched to the other drug which was continued for 30 days.
  Interventions: Drug: Atorvastatin; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Atorvastatin — Patients were randomly assigned to atorvastatin (40 mg day) for 30 days. After 1-week wash-out period to avoid any carryover effect, cross-over was performed, and patients were switched to the other drug which was continued for 30 days.
  Other Names: torvast, totalip
Drug: Rosuvastatin — Patients were randomly assigned to rosuvastatin (20 mg day) for 30 days. After 1-week wash-out period to avoid any carryover effect, cross-over was performed, and patients were switched to the other drug which was continued for 30 days.
  Other Names: crestor, provisacor,

SUMMARY:
Statin interference has been suggested among the mechanisms of reduction of the antiplatelet effect of clopidogrel. The purpose of this study is to evaluate pharmacodynamic effects of rosuvastatin and atorvastatin on platelet reactivity in patients with coronary artery disease undergone double antiplatelet therapy with new P2Y12 inhibitors. This is a single-center, prospective, randomized, crossover study conducted in the Department of Heart and Great Vessels "Attilio Reale", Sapienza University, Rome, Italy. All consecutive patients undergone PTCA in our institution in the period between July 2013 and December 2013 will be eligible to be enrolled.

Patients will be offered to participate to the trial at time of 1-month post-angioplasty follow-up visit.patients receiving dual antiplatelet therapy (prasugrel 10 mg or brilique 90 mg x 2 plus aspirin 100 mg) after percutaneous coronary intervention. Patients were randomly assigned to rosuvastatin (20 mg day) or atorvastatin (40 mg day) for 30 days. After 1-week wash-out period to avoid any carryover effect, cross-over was performed, and patients were switched to the other drug which was continued for 30 days.

Platelet function will be evaluated using a validated method: the VerifyNow System (Accumetrics Inc., San Diego, CA), which is a point-of-care turbidimetry-based optical detection system that measures platelet-induced aggregation. Platelet function will be measured with the VerifyNow P2Y12 test at baseline and after 30 days from rosuvastatin or atorvastatin administration.

Platelet reactivity will be expressed in P2Y12 reaction units (PRU). PRU values >208 are suggestive of high platelet reactivity.

DETAILED DESCRIPTION:
Statin interference has been suggested among the mechanisms of reduction of the antiplatelet effect of clopidogrel. The purpose of this study is to evaluate pharmacodynamic effects of rosuvastatin and atorvastatin on platelet reactivity in patients with coronary artery disease undergone double antiplatelet therapy with new P2Y12 inhibitors. This is a single-center, prospective, randomized, crossover study conducted in the Department of Heart and Great Vessels "Attilio Reale", Sapienza University, Rome, Italy.

ELIGIBILITY:
Inclusion Criteria:

1. Angiographically-proven coronary artery disease;
2. Able to understand and willing to sign the informed CF;
3. Stable clinical condition;
4. treatment with dual antiplatelet therapy (with P2Y12 inhibitors);

Exclusion Criteria:

1. Other drugs or medications that affect CYP mediated drug metabolism;
2. Allergy or adverse reactions to administered drugs;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of platelet reaction units | After 30 days of treatment with each drug
  Absolute changes in platelet reactivity (expressed as P2Y(12) reaction units by the point-of-care VerifyNow assay [Accumetrics, San Diego, California]

SECONDARY OUTCOMES:
Frequency of high platelet reactivity | After 30 days of treatment with each drug
  Frequency of high platelet reactivity with the 2 study treatments (as defined by a Platelet Reaction Unit value>208

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza Univeristy of Rome, Rome, Italy, Italy